CLINICAL TRIAL: NCT03208517
Title: An eLearning Optimized Person Centred Intervention to Improve Staff Attitudes and Quality of Care for People With Dementia Living in Care Homes
Brief Title: Improving Staff Attitudes and Care for People With Dementia: eLearning
Acronym: tEACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 196661 16/WA/0090 tEACH
Record Dates: First submitted 2017-06-29; First posted 2017-07-05 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2017-09

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Regular Contact Group (WHELD +) (Experimental): Regular Contact Group (WHELD elearning package + regular supervision support) A research associate will provide one face-to-face training session with participating care staff in the care home on how to use the online modules, providing a walk-through demonstration to ensure all are comfortable with the programme and its technology. The research associate will provide light touch support by returning fortnightly throughout the intervention period to the care home to observe/troubleshoot around online programme.
  Interventions: Other: Improving Wellbeing and Health for People with Dementia (WHELD) e-learning training programme
- Arm 2: Online Contact Group (WHELD only) (Experimental): Online Contact Group (WHELD elearning package only) The e-learning modules will be emailed to the care home with clearly written instructions on how to access the course.
  Interventions: Other: Improving Wellbeing and Health for People with Dementia (WHELD) e-learning training programme
- Arm 3: Enhanced usual practice Control Group (No Intervention): Arm 3: Enhanced usual practice Control Group (with information/signposting re high quality on line e-learning and educational materials).
  This will consist of a 2-page written guidance sheet on the best freely available dementia e-learning programmes and a one-off meeting with a research associate in the care home to explain the information/signposting

INTERVENTIONS:
Other: Improving Wellbeing and Health for People with Dementia (WHELD) e-learning training programme — The e-learning WHELD intervention The optimised e-learning programme will consist of five 25-minute interactive online modules based on a recently completed RCT of an in person training programme (WHELD), combining the most effective elements of existing approaches to create a comprehensive but practical staff training intervention. Based on a factorial study and qualitative evaluation, WHELD combines: person-centred care, person-centred activities and interactions, and updated knowledge regarding optimal use of psychotropic medications.
  Arms: Arm 1: Regular Contact Group (WHELD +); Arm 2: Online Contact Group (WHELD only)

SUMMARY:
The primary objective of this study is to determine whether a Person Centred Care online training programme confers significant benefit in terms of improving staff attitudes and quality of care of residents with dementia living in care homes, in comparison to enhanced usual training for professional care staff.

There is considerable interest in e-learning and dementia from care home providers. Significant investment has been made into the production of resources for care staff but to date there appears to be no, or very limited, evaluation of their effectiveness.

The aim is to provide a cost-effective, simple and practical evidence-based intervention, improving staff attitudes towards residents with dementia and quality of care provision. The trial will be a randomized controlled 3-arm cluster single blind trial that will take place over 9 months in 24 care homes in the UK.

DETAILED DESCRIPTION:
The National Institute for Health Research (NIHR) funded Well-being and Health for People with Dementia (WHELD) programme, An Optimized Person Centred Intervention to Improve Quality of Life for People with Dementia Living in Care Homes. This optimized intervention is based on a factorial study and qualitative evaluation, to combine: training on person-centred care, promoting person-centred activities and interactions, and providing care home staff and general practitioners with updated knowledge regarding optimal use of psychotropic medications for persons with dementia in care homes. Using a train-the-trainer model, the intervention was delivered by trained therapists, who trained 2 lead care staff members (WHELD champions) within each care home to implement the intervention over a 9-month period.

The primary objective of this study involving 24 care homes, with approximately 240 care staff, is to determine whether an online version of the optimized WHELD intervention, with or without supervision support, confers significant benefit in terms of improving attitudes of care staff caring for people with dementia and quality of care of residents with dementia living in care homes.

There is considerable interest in e-learning and dementia. Significant investment has been made into the production of resources for care staff but to date there appears to be no, or very limited, evaluation of the effectiveness of e-learning in either raising awareness amongst care staff, or increasing outcomes of care for people with dementia. In spite of the lack of evidence, e-learning remains popular with care home providers and managers, as they are perceived to be low-cost, can be delivered to staff on-site or even at home, and with minimal disruption to staffing routines and schedules.

The e-learning programme is based on the aforementioned WHELD RCT programme, which included over 80 care homes and 1000 participants in the study, and has already shown significant benefits in improvements in quality of life and agitation. This study will provide pilot testing to evaluate the effectiveness of an e-learning version.

Key secondary objectives will be to determine the specific impact of the e-learning intervention on a range of outcomes including quality of care, quality of the interaction of care staff with people with dementia, person-centered practice, staff knowledge about dementia and staff general health, work stress and experience working with residents with dementia.

The investigators hypothesize that the intervention (in particular with supervision support) will significantly improve several key outcomes. Specifically, the investigators hypothesize that, compared to enhanced usual training, the optimized e-learning intervention will:

• Improve staff attitudes towards people with dementia

The secondary hypotheses are that the WHELD e-learning intervention will:

* Improve quality of care
* Improve quality of interactions between staff and residents
* Improve person-centred practice
* Increase staff knowledge about dementia
* Improve staff general health
* Reduce staff work stress
* Improve satisfaction in caring for people with dementia

Baseline, post intervention and 4-month follow up data will be collected on all consented participants who meet the inclusion criteria at each participating care home.

ELIGIBILITY:
Care Home Selection:

Inclusion Criteria:

* Care homes that have residential or nursing status and are registered to provide care for people with dementia.
* Care homes randomly selected from the Care Home Research Network
* Research enabled and actively engaged in ENRICH programme
* Care homes should be able to demonstrate an acceptable standard of care according to Care Quality Commission (CQC).
* Prepared to release staff to complete training and to implement interventions
* Have a manager in post who is willing/able to act as key link person for trial
* "Tech ready" home - staff have access to PCs or tablets in the care home

Exclusion criteria:

* Less than 60% of the residents have dementia
* Care home is receiving special support from their local authority
* Care home has failed to meet more than 1 of the 5 CQC care home quality standards checks
* Insufficient staffing resource: Care home unable to provide care staff for training

Participant Selection:

Inclusion Criteria:

* Sufficient competence in English to undertake the training programme
* Qualified and unqualified paid care staff
* Permanent or contract employees providing direct care to residents
* Has basic computer literacy

Exclusion Criteria:

• Bank or agency staff

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Approaches to Dementia Questionnaire (ADQ) assessing change between time points | T1: baseline, T2: up to 2 weeks post intervention, T3: 4 month follow up
  This measure includes 19 attitudinal items, each scored from 1 (strongly disagree) to 5 (strongly agree) [3]. They are summed to form a total score (range 19-95) as well as a hope subscore (8 items, range 8-40) and a person-centred subscore (11 items, range 11-55). Higher scores indicate more positive attitudes. Example items indicative of hope (reverse scored) include ''people with dementia are very much like children'' and ''it is important not to become too attached to residents.'' Items related to person-centred care include ''it is important for people with dementia to be given as much choice as possible in their daily lives'' and ''people with dementia need to feel respected, just like anybody else.''

SECONDARY OUTCOMES:
Dementia Care Mapping assessing change between time points | T1: baseline, T2: up to 2 weeks post intervention, T3: 4 month follow up
  This measure will be used as an observation tool to assess quality of care [4]. DCM is an established and National Institute for Clinical Excellence/Social Care Institute for Excellence (NICE/SCIE) recommended, routine care home/NHS practice development intervention that is regularly used for ensuring a systematic approach to providing individualised person-centred care. It is used to support the sustained implementation of PCCT in dementia care practice. DCM is an observational tool, set within a practice development cycle. There is good evidence of its use in practice settings as a quality audit and improvement tool.
The General Health Questionnaire-12 assessing change between time points | T1: baseline, T2: up to 2 weeks post intervention, T3: 4 month follow up
  This measure is a widely used short screening instrument comprised of 12 items [5]. Goldberg and colleagues (1997) found the GHQ-12 to have good overall sensitivity (83.4%) and specificity (76.3%). The mean area under the ROC curves was 0.88 with a narrow range. Goldberg and colleagues (1997) scored the scales using both the GHQ method (0-0-1-1) as well as using a Likert method (0-1-2-3). It was found, for the GHQ-12, that the GHQ method was better for specificity and sensitivity than the Likert method. The GHQ-12's validity characteristics were not significantly different when accounting for gender, age group or educational level.
Staff Experience Working with Residents with Dementia assessing change between time points | T1: baseline, T2: up to 2 weeks post intervention, T3: 4 month follow up
  This measure includes 21 items assessing satisfaction, each scored from 0 (not at all) to 4 (extremely) and summed to create a total score ranging from 0 to 84 [6]. Higher scores indicate more satisfaction, and subscales can be created for each of six domains: (satisfaction with) feedback, the care organization, one's own expectations, patient contact, expectations of others, and the environment.
Knowledge in Dementia Scale assessing change between time points | T1: baseline, T2: up to 2 weeks post intervention, T3: 4 month follow up
  This measure is a 16-item self-report questionnaire used to measure knowledge in dementia [7]. The questionnaire is scored on an agree/disagree scale; 'agree' responses are given a score of 1, 'disagree' responses are given a score on 0. This means that it is possible to gain a total score between 0 and 16, a higher score being representative of better knowledge about dementia.
Quality of Interactions Schedule assessing change between time points | T1: baseline, T2: up to 2 weeks post intervention, T3: 4 month follow up
  This measure is an observational tool that measures the quality of interactions between staff and resident and person-centred environment in care home settings [8].
Inventory of Geriatric Nursing Self-Efficacy assessing change between time points | T1: baseline, T2: up to 2 weeks post intervention, T3: 4 month follow up
  This measure is a 9-item measure specifically developed for individuals providing nursing care to geriatric populations to quantify the extent to which individuals perceive themselves able to manage common sources of caregiver stress

CONTACTS AND LOCATIONS:
Overall Officials: Professor Clive Ballard, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided